CLINICAL TRIAL: NCT06305416
Title: Randomized, Double-blind, Parallel, Active Controlled Study to Compare Efficacy & Safety Between Ranibizumab 10mg/ml Injection of Incepta and Lucentis in Patients With Diabetic Macular Edema by ITV Injection
Brief Title: A Efficacy and Safety Study of Ranibizumab 10mg/ml Injection (Incepta) in Patients With Diabetic Macular Edema
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Incepta Pharmaceuticals Ltd (Industry)
Collaborators: Institute for Developing Science and Health Initiatives, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023/CT/01
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2024-11

CONDITIONS: Diabetic Macular Edema; Diabetic Retinopathy; Macular Edema; Macular Degeneration; Retinal Disease; Retinal Degeneration
Keywords: Ranibizumab; Efficacy; Diabetes; Retina; Edema
MeSH Terms: conditions — Diabetic Retinopathy; Macular Edema; Macular Degeneration; Retinal Diseases; Retinal Degeneration; Diabetes Mellitus; Edema | interventions — Ranibizumab; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ranibizumab 10mg/ml Injection (Proposed Ranibizumab Biosimilar) (Experimental): Test Group of 35 adult patient with DME will get Ranibizumab (Proposed Ranibizumab Biosimilar)
  Interventions: Drug: Ranibizumab 10mg/ml Injection
- Lucentis (Ranibizumab) (Active Comparator): Comparator Group of 35 adult patient with DME will get Lucentis
  Interventions: Drug: Lucentis

INTERVENTIONS:
Drug: Ranibizumab 10mg/ml Injection — Ranibizumab 10mg/ml Injection (proposed ranibizumab biosimilar) 0.5mg via intravitreal injection every 4 weeks
  Other Names: Test Product
  Arms: Ranibizumab 10mg/ml Injection (Proposed Ranibizumab Biosimilar)
Drug: Lucentis — Lucentis (ranibizumab) 0.5mg via intravitreal injection every 4 weeks
  Other Names: Reference Product
  Arms: Lucentis (Ranibizumab)

SUMMARY:
Macular edema in diabetes, defined as retinal thickening within two disc diameters of the center of the macula, results from retinal microvascular changes that compromise the blood-retinal barrier, causing leakage of plasma constituents into the surrounding retina and consequently retinal edema. Thickening of the basement membrane and reduction in the number of pericytes are believed to lead to increased permeability and incompetence of the retinal vasculature. This compromise of the blood-retinal barrier leads to the leakage of plasma constituents into the surrounding retina with subsequent retinal edema. Hypoxia produced by this mechanism can also stimulate the production of vascular endothelial growth factor (VEGF). Vascular endothelial growth factor (VEGF) increases retinal vascular permeability, causes breakdown of the blood-retina barrier and results in retinal edema.

Diabetic macular edema (DME) is the most common cause of visual reduction in patients with Diabetes Mellitus. The prevalence of DME globally is around 6.8 %. Diabetic Retinopathy (DR) is the most common microvascular complication of diabetes and the leading cause of blindness worldwide. DME is a complication of diabetic retinopathy that affects the macula, which is located at the center of the retina and responsible for central vision. Bangladesh is the 10th country in the world for the number of adults living with diabetes with some 7.1 million (5.3-12.0). In Bangladesh, it is therefore expected that diabetic secondary complications, like DR, will increase along with the rising trend of diabetes mellitus.

The use of therapeutic monoclonal antibodies has revolutionized in the treatment of many diseases. In recent years, millions of patients have been successfully treated with these biological agents. Ranibizumab is one such therapeutic monoclonal antibody for intraocular use. Ranibizumab is a humanized, recombinant, immunoglobulin G1 monoclonal antibody fragment against vascular endothelial growth factor A (VEGF-A) and thus prevents choroidal neovascularization. The small size of ranibizumab allows for enhanced diffusion into the retina and choroid.

DETAILED DESCRIPTION:
This is a randomized, double-blind, parallel study that will be conducted in patients with Diabetic Macular Edema (DME) to assess efficacy and safety between test and reference products. Total 70 subjects with DME are planned to be randomized into this study.

Enrolled subjects will receive total 3 doses of 0.5 mg Intravitreal injection of either test or reference product once every 4 Weeks (Day 0, Week 4±3 days and Week 8±3 days). All subjects will have their first injection of ranibizumab on Day 0 and undergo a safety visit 48hrs after the first injection. At subsequent visits, the subject will have a safety follow up prior to each intravitreal injection. Also the subject will have a safety follow up visit 48hrs after second and third injection. The final visit or end of study visit will be on Week 12±3 days for efficacy and safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Ages Eligible for Study: ≥ 18 Years
2. Ability to provide written informed consent and comply with study assessments for the full duration of the study
3. Diagnosis of diabetes mellitus (type 1 or 2). Any one of the following will be considered to be sufficient evidence that diabetes is present: Laboratory reports that prove DM of patient or current regular use of insulin for treatment of diabetes or current regular use of oral anti-hyperglycemic agent for the treatment of diabetes.
4. Clinical evidence of retinal thickening due to macular edema involving the center of the macula (can be associated with diabetic retinopathy)
5. Central diabetic macular edema present on clinical examination and OCT testing with central 1mm sub field thickness greater than 300 microns as measured on -OCT
6. Visual acuity score greater than or equal to 19 letters (20/400) and less than or equal to 73 letters (20/40) by the ETDRS/ Snellen chart visual acuity protocol
7. Media clarity, pupillary dilation and patient cooperation sufficient to allow OCT testing and retinal photography
8. Willingness and ability to undertake all scheduled visits and assessments

Exclusion Criteria:

1. Prior treatment with any Intravitreal drug, Bevacizumab, verteporfin or photodynamic therapy (except for extra foveal laser photocoagulation) in the study eye within past 3 months before study entry
2. Laser photocoagulation in the study eye within 1 month before study entry
3. Participation in another ocular investigation or trial simultaneously
4. Pregnancy (positive pregnancy test) or known to be pregnant; also pre-menopausal women not using adequate contraception.
5. Blood pressure > 160/100 mmHg (systolic above 160 or diastolic above 100) and Random Blood Sugar (RBS) ≥ 12 mmol/L and/ or HbA1c ≥ 7.5%
6. Evidence of vitreoretinal interface abnormality and optic nerve disease after ocular exam or OCT that may be contributing to the macular edema
7. Any concurrent intraocular condition in the study eye that could either require medical or surgical intervention during the study period or that could contribute to a loss of best corrected visual acuity over the study period (e.g. cataract that might decrease the vision by 3 or more lines, uncontrolled glaucoma, uveitis, previous corneal transplant etc.). The decision regarding exclusion is to be based on the opinion of the investigator.
8. An eye that, in the investigator's opinion, has no chance of improving in visual acuity following resolution of macular edema (e.g. presence of sub retinal fibrosis or geographic atrophy).
9. Presence of suspected ocular or periocular infections, another ocular condition that may affect the visual acuity or macular edema during the course of the study (uveitis, Irvine-Gas)
10. Vitreous hemorrhage preventing visualization of retina
11. History of vitreous surgery, cataract surgery, YAG capsulotomy in the study eye within last 3 months of enrolment
12. Visual acuity <20/400 in the fellow eye
13. Known hypersensitivity to Ranibizumab or any of the components of study medication
14. History of cerebral vascular accident or myocardial infarction within past 3 months.
15. Employees of Investigational sites, individuals directly involved with the conduct of the study or immediate family members thereof, prisoners, and persons who are legally institutionalized.
16. Current use of systemic medications known to be toxic to the lens, retina or optic nerve, including deferoxamine, chloroquine/ hydroxychloroquine, tamoxifen, phenothiazine, vigabatrin and ethambutol, and such medications will not be allowed during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-03-30 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Best Corrected Visual Acuity (BCVA) from Baseline | Baseline and Week 12
  To determine the changes in the BCVA was assessed using ETDRS charts or Snellen charts from baseline to Week 12
Changes in Central Subfield Thickness (CST) from Baseline | Baseline and Week 12
  To determine the changes in central 1mm subfield thickness as measured by OCT and FA from baseline to week 12

SECONDARY OUTCOMES:
Proportion of patients who lost fewer than 15 letters (approximately 3 lines) from baseline visual acuity | Baseline and Week 12
  The VA will be assessed using ETDRS charts or Snellen charts.
Proportion of patients who gained ≥15 letters (approximately 3 lines) from baseline visual acuity | Baseline and Week 12
  The VA will be assessed using ETDRS charts or Snellen charts.
Evaluation and comparison of safety between reference vs. test drug. | Baseline and upto Week 12
  Incidence of drug related adverse events as assessed by clinical and ophthalmic examination, vitals and laboratory parameters in both treatment arms

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Niaz Abdur Rahman, Principal Investigator — Managing Director, Bangladesh Eye Hospital & Institute
Locations (1):
- Bangladesh Eye Hospital & Institute, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
By publication in the journal
Supporting Information: Study Protocol, CSR
Time Frame: After completion of study
Access Criteria: Journal